CLINICAL TRIAL: NCT07112144
Title: Phase III Clinical Trials to Evaluate the Immunogenicity and Safety of Adsorption-free Diphtheria and Tetanus (Three-component) Combined Vaccine in 2-month-old Infants and Young Children
Brief Title: Adsorption of Cell-free Diphtheria and Tetanus (Three-component) Combined With Vaccine Phase III Clinical Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: Yunnan Provincial Center for Disease Control and Prevention (Unknown); Shaanxi Provincial Center for Disease Control and Prevention (Other); Guizhou Provincial Center for Disease Control and Prevention (Unknown); Shandong Provincial Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1004-F20240930-3
Record Dates: First submitted 2025-06-15; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Prevent Whooping Cough; Prevent Diphtheria; Prevent Tetanus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DTacP (Experimental)
  Interventions: Biological: DTacP
- DTaP (Active Comparator)
  Interventions: Biological: DTaP
- DTacP-IPV/Hib (Active Comparator)
  Interventions: Biological: DTacP-IPV/Hib

INTERVENTIONS:
Biological: DTacP — Vaccinate 1 dose at 2 months, 4 months, 6 months, 18-24 months and 6 years of age respectively, with each injection dose being 0.5 ml；Injection；
  Arms: DTacP
Biological: DTaP — Vaccinate 1 dose at 2 months, 4 months, 6 months, 18-24 months and 6 years of age respectively, with each injection dose being 0.5 ml.Injection
  Arms: DTaP
Biological: DTacP-IPV/Hib — Administer 1 dose at 2 months, 4 months, 6 months and 18 months of age respectively, with each injection dose being 0.5 ml.Injection
  Arms: DTacP-IPV/Hib

SUMMARY:
The immunogenicity and safety of the adsorption of cell-free diphtheria and tetanus (three-component) combined vaccine were evaluated at 2 months, 4 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants and young children who are permanent residents aged 2 months (60-89 days), and can provide valid identification documents for the subject and their legal guardian;
2. Obtain the informed consent of the subject's legal guardian and sign the informed consent form;
3. The legal guardian of the subject can comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

1. History of pertussis, diphtheria, or tetanus;
2. Contact with individuals diagnosed with pertussis or diphtheria within the past 30 days;
3. Vaccination with vaccines containing DTaP components, inactivated poliovirus vaccine, 13-valent pneumococcal polysaccharide conjugate vaccine, or Hib vaccine;
4. Premature infants (born before 37 weeks of gestation), infants with severe abnormal labor processes or a history of asphyxia rescue, or low birth weight infants (<2500g);
5. Axillary temperature >37.0°C on the day of enrollment*;
6. Severe congenital malformations or developmental disorders, genetic defects, severe malnutrition, or congenital diseases (such as Down syndrome, sickle cell anemia, congenital nervous system diseases, etc.);
7. History of epilepsy, convulsions, or seizures, history of cerebral palsy, or family history of mental illness;
8. Autoimmune diseases or immunodeficiencies (such as perianal abscesses suggesting possible immunodeficiency in infants, human immunodeficiency virus infection, lymphoma, leukemia, etc.), or parents/siblings with autoimmune diseases or immunodeficiencies;
9. Asplenia or splenic dysfunction due to any cause;
10. Clinically diagnosed coagulation disorders (such as coagulation factor deficiencies, coagulation diseases, platelet abnormalities) or obvious bruising/coagulation disorders that may contraindicate intramuscular injection;
11. History of severe allergic diseases (such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrotic reactions), history of severe allergic reactions to any vaccine (widespread urticaria, angioedema, etc.), or allergy to any known component of the test vaccine (pertussis toxoid, filamentous hemagglutinin, 69KD outer membrane protein, diphtheria toxoid, tetanus toxoid, aluminum hydroxide, sodium chloride, sodium hydroxide, etc.);
12. Vaccination with subunit or inactivated vaccines within the past 7 days; vaccination with live attenuated vaccines within the past 14 days*;
13. Receipt of immunoglobulin and/or any blood products (except hepatitis B immunoglobulin) before enrollment;
14. Receipt of any immunostimulant or immunosuppressant therapy before enrollment (continuous oral administration or infusion for ≥14 days, or topical steroid use [inhaled, nasal spray, intra-articular, eye drops, ointments, etc.] exceeding the recommended dosage in the package insert);
15. Suffering from acute illnesses within 3 days before enrollment (acute illness is defined as moderate or severe illness with or without fever)*;
16. Administration of prophylactic medications (such as antipyretic analgesics, antiallergic drugs, antidiarrheal drugs, etc.) within 3 days before enrollment*;
17. Known or suspected severe clinically diagnosed diseases (including but not limited to severe diseases of the nervous, cardiovascular, hematological and lymphatic, immune, renal, hepatic, gastrointestinal, respiratory, metabolic, and skeletal systems, as well as a history of malignant tumors);
18. Currently participating in other clinical trials or planning to participate in other trials during the study period;
19. Any other factors that, in the judgment of the researcher, make the subject unsuitable for participating in the clinical trial.

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1650 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | day 30 post-primary immunization
  The geometric mean concentration (GMC) of anti-PT antibody, anti-FHA antibody, anti-PRN antibody, anti-DT antibody, and anti-TT antibody at 30 days post-primary immunization
Immunogenicity | day 30 post-primary immunization
  Seroconversion rates of anti-PT, anti-FHA, anti-PRN, anti-DT, and anti-TT antibodies at day 30 post-primary immunization

SECONDARY OUTCOMES:
Immunogenicity | day 30 post-primary immunization
  Positivity rates of anti-PT, anti-FHA, anti-DT, and anti-TT antibodies at day 30 post-primary immunization
Immunogenicity | day 30 post-primary immunization
  Proportions of subjects with anti-PRN antibody levels ≥5, ≥10, and ≥20 IU/mL at day 30 post-primary immunization
Immunogenicity | day 30 post-fourth booster immunization
  Geometric mean concentrations (GMCs) of anti-PT, anti-FHA, anti-PRN, anti-DT, and anti-TT antibodies at day 30 post-fourth booster immunization
Immunogenicity | day 30 post-fourth booster immunization
  Seroconversion rates of anti-PT, anti-FHA, anti-PRN, anti-DT, and anti-TT antibodies at day 30 post-fourth booster immunization
Immunogenicity | day 30 post-fourth booster immunization
  Positivity rates of anti-PT, anti-FHA, anti-DT, and anti-TT antibodies at day 30 post-fourth booster immunization
Safety | At 12 months post-complete vaccination series
  Incidence of adverse events (AEs) and serious adverse events (SAEs) following each vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Yanshan County Center for Disease Control and Prevention, Wenshan Zhuang and Miao Autonomous Prefecture, Yunnan, China